CLINICAL TRIAL: NCT03454204
Title: Pharmacokinetic and Pharmacodynamic Modelling of Norepinephrine in Patients Under Target Controlled Infusions (TCI) for Anaesthesia : Plasma Concentration and "Site Effect"
Brief Title: Pharmacokinetic and Pharmacodynamic Modelling of Norepinephrine in Patients Under Target Controlled Infusions (TCI) for Anaesthesia
Acronym: NOR-PHARM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K170902J; 2017-A02671-52 (Other: IDRCB)
Record Dates: First submitted 2018-02-26; First posted 2018-03-05 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Neurosurgery; Intervention
MeSH Terms: interventions — Pharmacogenomic Variants

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pharmacokinetic: Establish a pharmacokinetic relationship between plasma concentration and the effect of norepinephrine in patients under concentration-target intravenous anesthesia by identifying significant covariates during general anesthesia.
  Interventions: Other: Pharmacokinetic

INTERVENTIONS:
Other: Pharmacokinetic — Analysis of blood samples

SUMMARY:
Currently, administration of norepinephrine diluted at 5 µg/ml bolus or continuous infusion is common during sympatholysis hypotension of TCI following the elimination of hypovolemia or anesthetic overdosage. Continued intravenous administration must meet hemodynamic goals within a narrow time frame. Depending on the intensity of hypotension the dosage is variable. It is adjusted in real time while it is excessive or insufficient at times. Therefore, the development of modeling should predict the kinetic and hemodynamic effects based on dosage and individual.

DETAILED DESCRIPTION:
Main objective Establish a pharmacokinetic relationship between plasma concentration and the effect of norepinephrine in patients under concentration-target intravenous anesthesia by identifying significant covariates during general anesthesia.

Primary Evaluation Criteria Relationship between exposure and the effect (desired-effectiveness or undesirable-toxicity) of norepinephrine during hypotension induced by anaesthetic drugs in a pharmacokinetic model (PLASMATIC DOSAGES) and pharmacodynamic model (HEMODYNAMIC EFFECTS MODELISED)

Experimental design This is a single-center, "non-interventional" study.

Population concerned The study involves major patients who have benefited from intraoperative hemodynamic optimization with norepinephrine (as noradrenaline tartrate) for maintaining blood pressure under general anaesthesia in neurosurgery and interventional neuroradiology in adults.

Research Proceedings Arterial catheter sampling for plasma noradrenaline assay

Individual benefit:

There is no benefit for the patient

Collective benefit:

Intraoperative hemodynamic optimization with the use of norepinephrine (as noradrenaline tartrate) to maintain blood pressure under general anaesthesia in neurosurgery and interventional neuroradiology in adults. Continued intravenous administration of norepinephrine should meet hemodynamic goals within a narrow time frame. Depending on the intensity of hypotension the dosage is variable. It is adjusted in real time while it is excessive or insufficient at times. Therefore, the development of modeling should predict the kinetic and hemodynamic effects based on dosage and individual.

Risks and minimal constraints added by the research No added risk This clinical research work is "non-interventional" on adult patients who benefit from a neurosurgical or neuroradiological intervention and whose blood pressure monitoring justifies the installation of a blood pressure catheter. The use of blood pressure monitoring and recording monitors and blood samples do not require any additional invasive procedures on patients since it uses the vascular accesses already in place.

The first sample (T0) is taken before the start of the infusion, thus determining the endogenous concentration (C0).

After a norepinephrine bolus, the second sample (T1) is taken at least 15 minutes after the start of the steady flow infusion or 10 minutes after the last flow change to measure the plateau concentration (C1) These fixed timeframes were calculated by taking into account an incompressible timeframe linked to the estimated dead catheter volume of 2 minutes plus the 5 half lives of norepinephrine estimated at 3-4 minutes.

A third sample (T2) is taken 10 minutes after a flow change or before the end of the infusion (end of the procedure).

To study the kinetics of the norepinephrine bolus, a rapid kinetics of 5 samples in TO, T30, T60, T120, T5 minutes is carried out in order to obtain the peak and speed of decrease in norepinephrine blood concentration for 5 patients.

Number of selected subjects Selection of patients up to 30 analysable patients Number of Centre : 1 Research Agenda inclusion period: 18 months duration of participation (treatment + follow-up): duration of the surgical intervention or interventional neuroradiology procedure: 1 day total duration: 18 months Number of planned inclusions by centre and month : 2 Number of subjects required : 30

Statistics

Descriptives: analysis by means of the two-step compartmental approach, which consists in estimating the pharmacokinetic parameters of each individual, then averaging them (obtaining the average pharmacokinetic parameters) and evaluating their distribution for the population studied.

Selection and incorporation of all significant covariates into the basic model by Ascending-descending strategy: the pre-selected covariates are tested one by one on the basic model. Those that meet the criteria described above are selected and introduced at the same time in the basic model. A descending construction is then carried out: the covariates are removed one by one. If the objective function does not increase by more than 6.63 points and the interindividual variability of the parameter of interest is not increased, the covariate is considered to be insignificant. This process is renewed until all covariates in the model are significant.

Validation of the model: Bayesian estimation: it allows once the final model has been validated, the estimation of pharmacokinetic or pharmacodynamic parameters for each individual by taking into account a priori the known information of fixed and random effects, population parameters, residual variability, the value of covariates of the different subjects and n observations of x subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patient > 18 years of age with neurosurgery or neurological interventional radiology for whom invasive monitoring of blood pressure is indicated.
* 2. Patient with persistent low blood pressure during the general anesthesia procedure (Fall > 30% of preoperative MAP registered after patient installation and/or MAP < 55 mmHg) and achieves the depth of anesthesia objective (BIS 40-50).

Exclusion Criteria:

* 1. A patient on a continuous infusion of norepinephrine or other catecholamine initiated in another department or facility or whose start was not recorded or whose dosage changes were unknown.
* 2. All causes of hypotension related to the patient's intervention or illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves major patients who have benefited from intraoperative hemodynamic optimization with norepinephrine (as noradrenaline tartrate) for maintaining blood pressure under general anaesthesia in neurosurgery and interventional neuroradiology in adults.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
PLASMATIC DOSAGES | 1 day
  Relationship between exposure and the effect (desired-effectiveness or undesirable-toxicity) of norepinephrine during hypotension induced by anaesthetic drugs in a pharmacokinetic model (PLASMATIC DOSAGES) and pharmacodynamic model (HEMODYNAMIC EFFECTS MODELISED)

CONTACTS AND LOCATIONS:
Overall Officials: Vallée Fabrice, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service Anesthésie-Réanimation - Hôpital Lariboisière, Paris, France

REFERENCES:
- [Background] Sun LY, Wijeysundera DN, Tait GA, Beattie WS. Association of intraoperative hypotension with acute kidney injury after elective noncardiac surgery. Anesthesiology. 2015 Sep;123(3):515-23. doi: 10.1097/ALN.0000000000000765. PMID 26181335
- [Background] Moerman AT, Vanbiervliet VM, Van Wesemael A, Bouchez SM, Wouters PF, De Hert SG. Assessment of Cerebral Autoregulation Patterns with Near-infrared Spectroscopy during Pharmacological-induced Pressure Changes. Anesthesiology. 2015 Aug;123(2):327-35. doi: 10.1097/ALN.0000000000000715. PMID 26035251
- [Derived] Kindermans M, Joachim J, Manquat E, Leve C, Hong A, Mateo J, Mebazaa A, Gayat E, De Backer D, Vallee F. Micro- and macrocirculatory effects of norepinephrine on anaesthesia-induced hypotension: a prospective preliminary study. BMC Anesthesiol. 2023 Nov 16;23(1):374. doi: 10.1186/s12871-023-02342-3. PMID 37974084